CLINICAL TRIAL: NCT03453385
Title: Clinical Outcomes of a Nationwide, Naturalistic E-Cig Trial (CONNECT)
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Matthew Carpenter, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 493; 1R01CA210625-01A1 (NIH)
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Smoking; Tobacco Use
Keywords: Smoking; Nicotine; Tobacco; Electronic Cigarette
MeSH Terms: conditions — Smoking; Tobacco Use; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will not receive an NJOY electronic cigarette to sample and will continue smoking their usual cigarettes as much or as little as they would like.
- Sampling (Experimental): Participants will receive an NJOY electronic cigarette to sample and will continue smoking their usual cigarettes as much or as little as they would like.
  Interventions: Behavioral: Electronic Cigarette

INTERVENTIONS:
Behavioral: Electronic Cigarette — An e-cigarette and four weeks of e-liquid provided to participants.
  Arms: Sampling

SUMMARY:
The purpose of this study is to measure changes in smoking behavior during and following sampling of an e-cigarette product. E-cigarettes are classified by the US Food and Drug Administration (FDA) as a tobacco product, though they contain no tobacco. Unlike regular cigarettes, which are burned (creating smoke that is inhaled), e-cigarettes include a heating element that vaporizes nicotine. E-cigarettes are likely much safer than conventional cigarettes, but they may not be entirely safe. We are testing the effects of one specific ecigarette (NJoy) on naturalistic changes in smoking behavior. Neither the tobacco industry nor any ecigarette manufacturer provides support of any kind to this study. There is no requirement to quit smoking in this study, nor is there any requirement to use e-cigarettes.

DETAILED DESCRIPTION:
Eligible smokers, once consented, will be randomized to receive a sample of ecigarettes (NJoy Pre-Filled Tank; n=440) or not (n=220). E-cigarette samples are inclusive of a battery and self-contained tanks of assorted flavors to last up to 4 weeks. Participants will be recruited nationally, but a subset (N=120) will be recruited locally to allow for biomarker collection . Our two-fold purpose is to 1) characterize naturalistic uptake of e-cigarettes, and 2) assess impact of e-cigarette uptake on smoking behavior. All smokers will be asked to provide smoking diary data, captured electronically, daily for 4 weeks. More substantive phone assessment will track smoking and related behaviors at baseline (Day 0) and +10, +17, and +24 days (weekly during initial 3 weeks, following brief lag for delays in product mailing), and at +1, +3, and +6 months.

ELIGIBILITY:
Inclusion Criteria:

* age 21+,
* current smoker
* regular use of email OR capacity to receive SMS text and internet access
* additional smoking and health criteria determined at screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carpenter MJ, Wahlquist AE, Dahne J, Gray KM, Cummings KM, Warren G, Wagener TL, Goniewicz ML, Smith TT. Effect of unguided e-cigarette provision on uptake, use, and smoking cessation among adults who smoke in the USA: a naturalistic, randomised, controlled clinical trial. EClinicalMedicine. 2023 Aug 15;63:102142. doi: 10.1016/j.eclinm.2023.102142. eCollection 2023 Sep. PMID 37753443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Sampling
Started | 211 | 427
Completed | 211 | 427
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Sampling | Total
Number analyzed (Participants) | 211 | 427 | 638
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (11.9) | 42.4 (11.2) | 42.2 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 222 | 342
  Male | 91 | 205 | 296
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 63 | 90
  Not Hispanic or Latino | 184 | 364 | 548
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 146 | 291 | 437
  Black | 32 | 86 | 118
  Other | 33 | 50 | 83
Motivation to Quit Smoking (0-10 scale) [Mean (Standard Deviation); unit: units on a scale] — 0 is the lowest motivation and 10 is the highest motivation
  units on a scale | 4.5 (3.1) | 4.3 (3.3) | 4.4 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: E-cig Use at End of Sampling Period
Description: percentage of participants reporting using an e-cigarette
Time Frame: at week 4
Measure: Number; unit: percentage of participants
Arm/Group | Control | Sampling
Number analyzed (Participants) | 211 | 427
percentage of participants | 13 | 72

2. Secondary Outcome: Conversion
Description: Percentage of participants who purchase an e-cigarette or additional nicotine liquid on their own
Time Frame: Study enrollment through end of 6-month follow up
Measure: Number; unit: percentage of participants
Arm/Group | Control | Sampling
Number analyzed (Participants) | 211 | 427
percentage of participants | 20 | 19

3. Secondary Outcome: Smoking Cessation
Description: Point prevalence abstinence from conventional smoking
Time Frame: at 6-month follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Control | Sampling
Number analyzed (Participants) | 211 | 427
percentage of participants | 8 | 14

ADVERSE EVENTS:
Time Frame: study weeks 1 through 24
Description: AEs are asked of both groups at follow-up calls at Weeks 1, 2, 3, 4, 12, and 24.
Arm/Group | Control | Sampling
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/427
Serious Adverse Events (participants affected / at risk) | 0/211 | 1/427
Other Adverse Events (participants affected / at risk) | 98/211 | 177/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=211) | Sampling (N=427)
asthma-induced hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=211) | Sampling (N=427)
cough (Respiratory, thoracic and mediastinal disorders) | 43 | 73
headache (Nervous system disorders) | 17 | 52
increased phlegm (Gastrointestinal disorders) | 38 | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03453385/Prot_SAP_000.pdf